CLINICAL TRIAL: NCT02283229
Title: Newborn Head Molding and Later Asymmetries in Follow up (3D Head Shape Modelling)
Brief Title: Newborn Head Molding and Later Asymmetries
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Marita Valkama, PhD, M.D. Adjunct Professor, pediatrician and neonatologist, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EETTMK:27/2011
Record Dates: First submitted 2014-10-28; First posted 2014-11-05 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Plagiocephaly
Keywords: Plagiocephaly; torticollis; occlusal defect
MeSH Terms: conditions — Plagiocephaly; Torticollis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): Newborns with preventive caring advices
  Interventions: Behavioral: Newborns with preventive caring advices
- Surveillance (Placebo Comparator): Newborns with normal caring advices
  Interventions: Other: Newborns with normal caring advices

INTERVENTIONS:
Behavioral: Newborns with preventive caring advices — Advices to prevent head molding
  Arms: Active
Other: Newborns with normal caring advices — Normal handling
  Arms: Surveillance

SUMMARY:
Prospective randomized clinical interventional trial after birth in maternity ward, and follow up to 8-9 years of age.

Hypothesis: Preventive handling and caring advices to parents of newborns decrease craniofacial asymmetries (deformational plagiocephaly and torticollis). The minimum sample size of the study was calculated at 86 (43 in each arm) using a 5% significance level, a power of 80% and a fall in the prevalence of DP from 31% to 8%. Craniofacial asymmetries and appearances of occlusal defects are followed up to 9 years. 50 preterm infants can participate without intervention.

DETAILED DESCRIPTION:
The amount of craniofacial abnormal molding after birth in newborns and the frequency of plagiocephaly in infancy or later consequences of those in childhood are not known in finnish population. Head malposition and deformational plagiocephaly, however, have been linked to delayed development in early life and even much later to orthognathic problems demanding surgery in adulthood.

In this study parents with healthy newborns are randomized to have normal discharge home or discharged with extra advice information for caregivers; to charge both sided feeding and handling habits; to change regularly sleeping and lying positions; to have early tummy times.

Anthropometric measurements of the infants; tilting degrees of the head and rotations of the neck (range of movement =ROM) are taken at discharge home and at the age of 3 and 6 months, and 1, 3, 5-6 and 8-9 years. Two-dimensional digital photographs (upto the age of 6 months) and three-dimensional imaging (from the age of 3 months) are taken to measurements of the head shape (Cephalic index=CI and (approximate) Oblique Cranial Length Ratio= (a)OCLR measured using a semiautomated, computer-based method). The development quotient by Griffiths scales are assessed at the age of 3 and 6 months. Dental occlusal defect evaluation are started at the age of 3 ys.

ELIGIBILITY:
Inclusion Criteria:

* 1-6 days after birth;
* Healthy newborns in maternal ward, and living in near by Oulu region.
* Preterms at the age of 34-44 gestation weeks in near by Oulu region (non randomized)

Exclusion Criteria:

* Congenital anomalies,
* Very early discharge,
* Parental refusal

Ages: 1 Day to 6 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 135 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Presence of Plagiocephaly (The number of children in groups with plagiocephaly (CI, OCLR =/> 104% ) | 3 months
  The number of children in groups with plagiocephaly (CI, OCLR =/> 104%)

SECONDARY OUTCOMES:
Severity of plagiocephaly | 3 months
  The number of children in groups with plagiocephaly as mild; aOCLR 104-107%; moderate 107-111%; severe =/>111 %
Change in plagiocephaly | From 3 to 6 months
  The number of children in groups with plagiocephaly as mild; aOCLR 104-107%; moderate 107-111%; severe =/>111 %
Occlusal defects | 6 years
  The number of children in groups with occlusal defects
Change in occlusal defects | from 6 years to 10 years
  The number of children with occlusal defects
Change in facial symmetry | from 6 years to 10 years
  The number of children with facial asymmetry
Change in occlusal defects | from 10 years to 15 years
  The number of children with occlusal defects
Change in facial symmetry | from 10 years to 15 years
  The number of children with facial asymmetry

OTHER OUTCOMES:
Development (Development quotients by Griffiths scales in groups) | 3 months
  Difference in Development quotients by Griffiths scales in groups
Change in Development (Development quotients by Griffiths scales in groups) | From 3 months to 6 months
  Difference in Development quotients by Griffiths scales in groups

CONTACTS AND LOCATIONS:
Overall Officials: Pertti Pirttiniemi, Professor, Study Chair — University of Oulu; Marita Valkama, Ph.D., M.D., Principal Investigator — University of Oulu, Oulu University Hospital; Virpi Harila, Ph.D., Study Director — University of Oulu; Henri Aarnivala, M.D., Principal Investigator — University of Oulu; Tuomo Heikkinen, Dos, Principal Investigator — University of Oulu; Ville Vuollo, Ph.M., Principal Investigator — University of Oulu
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aarnivala HE, Valkama AM, Pirttiniemi PM. Cranial shape, size and cervical motion in normal newborns. Early Hum Dev. 2014 Aug;90(8):425-30. doi: 10.1016/j.earlhumdev.2014.05.007. Epub 2014 Jun 13. PMID 24951081
- [Result] Aarnivala H, Vuollo V, Harila V, Heikkinen T, Pirttiniemi P, Valkama AM. Preventing deformational plagiocephaly through parent guidance: a randomized, controlled trial. Eur J Pediatr. 2015 Sep;174(9):1197-208. doi: 10.1007/s00431-015-2520-x. Epub 2015 Apr 1. PMID 25823758
- [Result] Vuollo V, Holmstrom L, Aarnivala H, Harila V, Heikkinen T, Pirttiniemi P, Valkama AM. Analyzing infant head flatness and asymmetry using kernel density estimation of directional surface data from a craniofacial 3D model. Stat Med. 2016 Nov 20;35(26):4891-4904. doi: 10.1002/sim.7032. Epub 2016 Jul 6. PMID 27383684
- [Result] Aarnivala H, Vuollo V, Harila V, Heikkinen T, Pirttiniemi P, Holmstrom L, Valkama AM. The course of positional cranial deformation from 3 to 12 months of age and associated risk factors: a follow-up with 3D imaging. Eur J Pediatr. 2016 Dec;175(12):1893-1903. doi: 10.1007/s00431-016-2773-z. Epub 2016 Sep 13. PMID 27624627
- [Result] Launonen AM, Vuollo V, Aarnivala H, Heikkinen T, Pirttiniemi P, Valkama AM, Harila V. Craniofacial Asymmetry from One to Three Years of Age: A Prospective Cohort Study with 3D Imaging. J Clin Med. 2019 Dec 27;9(1):70. doi: 10.3390/jcm9010070. PMID 31892114
- [Result] Launonen AM, Aarnivala H, Kyteas P, Vuollo V, Heikkinen T, Kau CH, Pirttiniemi P, Harila V, Valkama AM. A 3D Follow-Up Study of Cranial Asymmetry from Early Infancy to Toddler Age after Preterm versus Term Birth. J Clin Med. 2019 Oct 11;8(10):1665. doi: 10.3390/jcm8101665. PMID 31614700